CLINICAL TRIAL: NCT03106428
Title: A Phase 1 Multicenter, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Antitumor Activity of MEDI7247 in Patients With Selected Relapsed/Refractory Hematological Malignancies
Brief Title: A Multiple Ascending Dose Study of MEDI7247 in Patients With Selected Relapsed/Refractory Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8540C00001
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia; Multiple Myeloma; Diffuse Large B-cell Lymphoma
Keywords: MEDI7247; Acute Myeloid Leukemia; Multiple Myeloma; Diffuse Large B-cell Lymphoma; AML; MM; DLBCL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- acute myeloid leukemia (Experimental): Patients with R/R AML by World Health Organization (WHO) classification (Arber et al, 2016) who have failed prior standard therapy and for whom no standard therapies are available
  Interventions: Drug: MEDI7247
- Multiple Myeloma (Experimental): Patients with R/R MM who have failed prior standard therapy(ies) which should include immunomodulatory agents and proteasome inhibitors and for whom there is no standard salvage regimen.
  Interventions: Drug: MEDI7247
- Diffuse Large B-cell Lymphoma (Experimental): Patients with R/R DLBCL who have failed prior standard therapy(ies) and for whom there is no standard salvage regimen.
  Interventions: Drug: MEDI7247

INTERVENTIONS:
Drug: MEDI7247 — The study will enroll patients with R/R AML/MM/DLBCL who will receive MEDI7247 IV

SUMMARY:
To assess safety and tolerability, describe the dose-limiting toxicities, determine the maximum tolerated dose (MTD) or the highest protocol-defined dose (maximum administered dose) in the absence of establishing the MTD, and a recommended dose for further evaluation of MEDI7247 in patients with selected hematological malignancies who have relapsed after, or are refractory to prior standard therapy, and for whom there is no standard salvage regimen available.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed relapsed/refractory diagnosis of select hematologic malignancies for which no standard/salvage therapies are available.
2. Age ≥ 18 years at the time of screening.
3. Written informed consent and any locally required authorization
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Liver Function Tests: AST and ALT ≤ 3 × ULN, and serum TBL ≤ 1.5 × ULN, unless consistent with Gilbert's syndrome for which TBL ≤ 2.5 × ULN is allowed.

5. CrCL ≥ 40 mL/min 6. Female patients of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception from 7 days post-screening, and must agree to continue using such precautions for 90 days after the last dose of investigational product.

7. Nonsterilized male patients who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide from 7 days post-screening and for 90 days after receipt of the last dose of investigational product.

Exclusion Criteria:

1. Received cytotoxic chemotherapy within 21 days (or 42 days for nitrosureas or mitomycin C) prior to the first scheduled dose of MEDI7247.
2. Received major surgery (as defined by the Investigator), radiotherapy, or immunotherapy (including immune checkpoint inhibitors and adoptive cellular therapy such as autologous or donor NK cell or T lymphocyte infusions (e.g. CAR -T cells)) within 28 days of the first scheduled dose of MEDI7247.
3. Received an investigational drug within 14 days of the first scheduled dose of MEDI7247 or not recovered from associated toxicities.
4. Patients who have previously received an autologous SCT, are excluded if less than 120 days have elapsed from the time of transplant or the patient has not recovered from transplant-associated toxicities prior to the first scheduled dose of MEDI7247.
5. History of liver cirrhosis, liver fibrosis or prior liver irradiation regardless of the time interval (not including total body irradiation administered during allogeneic SCT).
6. Failure to recover from all prior treatment-related non-hematological toxicities to ≤ Grade 1 prior to the first scheduled dose of MEDI7247 (except for alopecia and neuropathy).
7. Patients at risk of non-disease related major bleeding (eg, recent GI hemorrhage or neurosurgery, within previous 21 days).
8. Current severe active systemic disease including active concurrent malignancy
9. Central nervous system (CNS) disease that is untreated, symptomatic, or requires therapy to control symptoms.
10. Active human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infections at the time of screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) | From time of informed consent through 90 days post end of treatment
  To assess by the occurrence of adverse events (AEs)
Occurrence of serious adverse events (SAEs) | From time of informed consent through 90 days post end of treatment
  To assess by the occurrence of serious adverse events (SAEs)
Occurrence of dose-limiting toxicities (DLTs) | During the evaluation period of 21 or 42 days post-first dose
  To assess by the occurrence of non-Hematologic and hematologic toxicities, AEs, and abnormal laboratory results.
Number of patients with changes in laboratory parameters from baseline | From time of informed consent and up to 21 days post end of treatment
  To assess serum chemistry, hematology, Coagulation and urinalysis
Number of patients with changes in vital signs from baseline | From time of informed consent and up to 21 days post end of treatment
  To assess body temperature, blood pressure, and heart rate
Number of patients with changes in electrocardiogram (ECG) results from baseline | From time of informed consent and up to 21 days post end of treatment
  To assess using twelve-lead ECG recordings
Percentage of patients with changes in laboratory parameters from baseline | From time of informed consent and up to 21 days post end of treatment
  To assess serum chemistry, hematology, Coagulation and urinalysis

SECONDARY OUTCOMES:
MEDI7247 maximum observed concentration for PK | From time of informed consent through 30 days post end of treatment
  To assess the Pharmacokinetics of MEDI7247
MEDI7247 area under the concentration-time curve for PK | From time of informed consent through 30 days post end of treatment
  To assess the Pharmacokinetics of MEDI7247
MEDI7247 clearance for PK | From time of informed consent through 30 days post end of treatment
  To assess the Pharmacokinetics of MEDI7247
MEDI7247 terminal half-life for PK | From time of informed consent through 30 days post end of treatment
  To assess the Pharmacokinetics of MEDI7247
Number of subjects who develop anti-drug antibodies (ADAs) | From time of informed consent through 30 days post end of treatment
  To assess the immunogenicity of MEDI7247
Best overall response (BOR) | From time of informed consent and up to 3 years after final patient is enrolled
  To assess the anti-tumor activity of MEDI7247
Objective response rate (ORR) | From time of informed consent and up to 3 years after final patient is enrolled
  To assess the anti-tumor activity of MEDI7247
Time to response (TTR) | From time of informed consent and up to 3 years after final patient is enrolled
  To assess the anti-tumor activity of MEDI7247
Duration of response (DoR) | From time of informed consent and up to 3 years after final patient is enrolled
  To assess the anti-tumor activity of MEDI7247
Progression-free survival (PFS) | From time of informed consent and up to 3 years after final patient is enrolled
  To assess the anti-tumor activity of MEDI7247
Overall survival (OS) | From time of informed consent and up to 3 years after final patient is enrolled
  To assess the anti-tumor activity of MEDI7247

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Research Site, Los Angeles, California
  - Research Site, Denver, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Greer, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
- France (2):
  - Research Site, Pierre-Bénite
  - Research Site, Villejuif
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maris M, Salles G, Kim WS, Kim TM, Lyons RM, Arellano M, Karmali R, Schiller G, Cull E, Abboud CN, Batlevi C, Kagiampakis I, Rebelatto MC, Lee Y, Kirby LC, Wang F, Bothos J, Townsley DM, Fathi AT, Ribrag V. ASCT2-Targeting Antibody-Drug Conjugate MEDI7247 in Adult Patients with Relapsed/Refractory Hematological Malignancies: A First-in-Human, Phase 1 Study. Target Oncol. 2024 May;19(3):321-332. doi: 10.1007/s11523-024-01054-z. Epub 2024 Apr 29. PMID 38683495